CLINICAL TRIAL: NCT03014960
Title: The Effects of Leader Sleep Improvement on Leadership
Brief Title: Effects of Leader Sleep Improvement on Leadership
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Yu Tse Heng, Doctoral Student, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00000461-B
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Insomnia, Primary; Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Condition (Experimental): Online Cognitive Behavioral Therapy for Insomnia Intervention
  Interventions: Other: Online Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Control Condition (No Intervention): No intervention

INTERVENTIONS:
Other: Online Cognitive Behavioral Therapy for Insomnia (CBT-I) — CBT-I is a psychological treatment designed to break the patterns of maladaptive thinking and behavior that maintain insomnia. CBT-I includes a range of techniques including a behavioral component (stimulus control, sleep restriction, relaxation) combined with a cognitive component (managing sleep related worries, the racing mind and intrusive thoughts) and an educational (sleep hygiene) component.
  Arms: Experimental Condition

SUMMARY:
The purpose of the study is to investigate the effects of sleep improvement in leaders on leader outcomes.

DETAILED DESCRIPTION:
The investigators seek to extend the findings of a recent research which demonstrated that treating insomnia has several beneficial effects on employee work outcomes (Barnes, Miller, & Bostock, in press). In the present study, the investigators propose that the treatment of leader insomnia would beneficially influence leadership, specifically abusive supervision, charismatic leadership, and laissez-faire leadership.

ELIGIBILITY:
Inclusion criteria:

* Working adults who have at least one direct report (i.e., subordinate).

Exclusion criteria:

* Non-working adults/ adults who do not have at least one direct report (i.e., subordinate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Self-Control Scale | 2 weeks
  Rate self-control over the past 2 weeks. Each item is scored 1-5 (1 = Very slightly or not at all, 2 = A little, 3 = Moderately, 4 = Quite a bit, 5 = Extremely).
Abusive Supervision Scale | 2 weeks
  Rate abusive supervision over the past 2 weeks. Each item is scored 1-5:
  1. - I cannot remember him/her ever using this behavior with me
  2. - He/she very seldom uses this behavior with me
  3. - He/she occasionally uses this behavior with me
  4. - He/she uses this behavior moderately often with me
  5. - He/she uses this behavior very often with me
Emotional Labor Scale | 2 weeks
  Rate emotional labor over the past 2 weeks. Each item is scored 1-5 (1 = Very slightly or not at all, 2 = A little, 3 = Moderately, 4 = Quite a bit, 5 = Extremely).
Charismatic Leadership Scale | 2 weeks
  Rate charismatic leadership over the past 2 weeks. Each item is scored 1-5 (1 = to a very little extent; 2 = to a little extent; 3 = to a moderate extent; 4 = to a great extent; 5 = to a very great extent).
Emotional Exhaustion Scale | 2 weeks
  Rate emotional exhaustion over the past 2 weeks. Each item is scored 1-5 (1 = Very slightly or not at all, 2 = A little, 3 = Moderately, 4 = Quite a bit, 5 = Extremely).
Laissez-Faire Leadership Scale | 2 weeks
  Rate laissez-faire leadership over the past 2 weeks. Each item is scored 1-5 (1 = to a very little extent; 2 = to a little extent; 3 = to a moderate extent; 4 = to a great extent; 5 = to a very great extent).

SECONDARY OUTCOMES:
Insomnia Scale | 2 weeks
  Rate insomnia over the past 2 weeks. Each item is scored 1-5 (1 = Very slightly or not at all, 2 = A little, 3 = Moderately, 4 = Quite a bit, 5 = Very much)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Tse Heng, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No